CLINICAL TRIAL: NCT04359537
Title: Comparative Efficacy of Various Doses of Hydroxychloroquine in Pre-Exposure Prophylaxis for COVID 19 in Healthcare Personnel
Brief Title: Efficacy of Various Doses of Hydroxychloroquine in Pre-Exposure Prophylaxis for COVID 19
Acronym: CHEER
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Responsible Party: Principal Investigator, Fibhaa Syed, Assistan Professor Medicine, Shaheed Zulfiqar Ali Bhutto Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: F.1-1/2015/ERB/SZABMU/549
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: COVID 19
Keywords: pre-exposure prophylaxis; Healthcare personnel
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Participants fulfilling the eligibility criteria will be randomized to 4 arms by using Random Allocation Software version-2
  Arm Intervention /treatment Experimental group 1: Hydroxychloroquine 400 mg twice a day 1,followed by 400 mg weekly for a total of 12 weeks
  Experimental group 2:Hydroxychloroquine 400 mg on day 1 followed by 400 mg once every 3 weeks for a total of 12 weeks
  Experimental group 3:Hydroxychloroquine 200 mg on day 1 followed by 200 mg once every 3 weeks for a total of 12 weeks
  Control Group :Placebo 200mg will be given on day 1 followed by Placebo 200mg every three weeks for a total of 12 weeks..
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1 (Experimental): Hydroxychloroquine Sulphate will be administered at a dose of 400mg twice a day on day 1 followed by 400 mg once a week for a total of 12 weeks
  Interventions: Drug: Hydroxychloroquine Sulfate 200 MG
- Arm 2 (Experimental): Hydroxychloroquine Sulphate will be admoinistered at a dose of 400 mg on day 1 followed by 400mg once every 3 weeks for at total of 12 weeks
  Interventions: Drug: Hydroxychloroquine Sulfate 200 MG
- Arm 3 (Experimental): Hydroxychloroquine Sulphate will be administered at a dose of 200 mg on day 1 followed by 200 mg once every 3 weeks for a total of 12 weeks
  Interventions: Drug: Hydroxychloroquine Sulfate 200 MG
- Arm 4 (Placebo Comparator): Control group will recieve Placebo 200mg on day 1 followed by Placebo 200mg every three weeks for 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine Sulfate 200 MG — Hydroxychloroquine Sulphate 200 mg tablets will be prescribed and instituted orally at the doses and regimens described
  Other Names: Tab HCQ
  Arms: Arm 1; Arm 2; Arm 3
Other: Placebo — Control group will receive a Placebo tablet. Placebo 200mg will be given on Day 1 followed by Placebo 200mg every three weeks.
  Arms: Arm 4

SUMMARY:
Hydroxychloroquine has been approved by FDA as one of the treatment options for COVID 19.Healthcare personnel are amongst those at highest risk to contract the disease. Several health authorities are now recommending the use of hydroxychloroquine as pre-exposure prophylaxis is in health care personnel. Several studies are on going in this context. However there is a controversy regarding the dosage regimen. This drug has a half life of 22.4 days. In this study we will be comparing three different doses of Hydroxychloroquine and additionally have a control group in order to determine the efficacy of hydroxychloroquine as pre- exposure prophylaxis in healthcare personnel in various doses.

DETAILED DESCRIPTION:
Study design:

Phase 2 proof of concept study Study Type: Interventional (Clinical Trial) Estimated Enrollment : at least 200 participants Since the investigators have no current data on pre-exposure prophylaxis to calculate sample size statistically, so a minimum of 50 participants in each arm will be recruited including 20% attrition rate. The investigators will be recruiting a minimum of 200 participants in the study , that is at least 50 in each of the four arms.

Allocation: Randomized Intervention Model: Parallel Assignment Study model: Parallel group interventional study Location: SZABMU/PIMS Study duration: a minimum of 12 weeks from recruitment

Materials and Methods:

Participants will be recruited after approval from Ethical Review Board .A written informed consent will be taken from all participants. Participants fulfilling the eligibility criteria will be randomized to 4 arms.

Arm Intervention /treatment

Experimental group 1: Hydroxychloroquine 400 mg twice a day 1,followed by 400 mg weekly for a total of 12 weeks Drug: Hydroxychloroquin HCQ 200 mg, oral

Experimental group 2:Hydroxychloroquine 400 mg on day 1 followed by 400mg once every 3 weeks for a total of 12 weeks Drug: Hydroxychloroquin HCQ 200 mg, oral

Experimental group 3:Hydroxychloroquine 200 mg on day 1 followed by 200 mg once every 3 weeks for a total of 12 weeks Drug: Hydroxychloroquin HCQ 200 mg, oral

Control Group : Placebo 200mg will be given on day 1 followed by Placebo 200mg every three weeks for a total of 12 weeks.

Base line characteristics of all participants will be recorded including age ,gender,role of healthcare personnel, comorbidities, and drugs the participant is using.

Samples will be collected for complete picture blood, liver and renal function tests and electrocardiogram. These tests will also be conducted every month till the end of the trial and the participants will be monitored for any adverse effects.

During the study duration all participants will self- report any symptoms related to COVID 19 and any adverse reactions from the drug. Participants having COVID 19 symptoms at any time will be tested by the gold standard test PCR for SARS-COV-2 using nasopharyngeal and oropharyngeal swabs.

All participants at the end of the study will have PCR for SARS-COV-2 and if available IgM and IgG serology to find out if they had any infection, did not get infected at all or only had asymptomatic or mild infection.

ELIGIBILITY:
Inclusion Criteria after taking a written informed consent:

* A healthcare worker at high risk for COVID19 exposure (defined below):

  * Persons primarily working in emergency departments (physicians, nurses, ancillary staff, triage personnel) ;
  * Persons primarily working in intensive care units (physicians, nurses, ancillary staff, respiratory therapists) ;
  * Persons performing aerosol generating procedures (i.e. anesthesiologists, nurse anesthetists, gastroenterologists performing endoscopy, Pulmonologists performing bronchoscopy);
  * First responders (i.e. EMTs, paramedics) ;
  * Persons working in the departments of General Medicine, Pulmonology, Infectious disease and Isolation wards.

Exclusion Criteria:

* Active COVID-19 disease;
* Confirmed prior COVID-19 disease;
* Current fever, cough, shortness of breath;
* Contraindication or hypersensitivity to chloroquine or hydroxychloroquine ad hypersensitivity to 4-aminoquinoline compounds;
* Pregnancy;
* Lactation;
* Prior retinal eye disease;
* Known Chronic Kidney disease, Stage 4 or 5 or dialysis;
* Known glucose-6 phosphate dehydrogenase (G-6-PD) deficiency ;
* Weight <40 kg;
* Current use of chloroquine,hydroxychloroquine or cardiac medicines like flecainide, amiodarone, digoxin, procainamide, or propafenone;
* Current use of medications with known significant drug-drug interactions: artemether, lumefantrine, mefloquine, tamoxifen or methotrexate;
* Current use of medications causing QT interval prolongation like: macrolides,antipsychotics,quinolones,antihistamines,SSRIs,tricyclic antidepressants, antifungals;
* Recent Myocardial Infarction;
* History of Epilepsy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-08-25 (Estimated); Study Completion 2020-09-25 (Estimated)

PRIMARY OUTCOMES:
COVID-19-free survival in experimental arms compared to placebo | 12 weeks
  Outcome reported as the percentage of participants in each arm who are COVID-19-free at the end of study treatment

SECONDARY OUTCOMES:
Incidence of confirmed SARS-COV-2 detection | 12 weeks
  Outcome reported as the percent of participants in each arm who have a confirmed SARS-CoV-2 infection during study treatment.
Incidence of possible COVID-19 symptoms | 12 weeks
  Outcome reported as the percent of participants in each arm who report COVID-19-related symptoms during study treatment
Incidence of all-cause study medicine discontinuation | 12 weeks
  Outcome reported as the percent of participants in each arm who discontinue study medication use for any reason during treatment.
Ordinal Scale of COVID-19 Disease maximum severity if COVID-19 diagnosed at study end | 12 weeks
  Participants will self-report COVID-19 status on an ordinal scale as follows: No illness (score=1), Illness with outpatient observation (score=2), Hospitalization (or post-hospital discharge) (score=3), Hospitalization with ICU stay (score 4),Death from COVID 19(score=5) Possible scores range from 1-5 with higher scores indicating greater disease severity.
Incidence of Hospitalization for COVID-19 or death | 12 weeks
  Outcome reported as the percent of participants in each arm who are hospitalized or expire due to COVID-19 during study treatment.
Incidence of study medication-related adverse events | 12 weeks
  Outcome reported as the percent of participants experiencing any possible adverse events from Hydroxychloroquine

CONTACTS AND LOCATIONS:
Overall Officials: Fibhaa Syed, FRCP, Principal Investigator — Shaheed Zylfiqar Ali Bhutto Medical University; Mohammed Ali Arif, FRCP, Principal Investigator — Shaheed Zulfiqar Ali Bhutto Medical University; Rauf Niazi, FRCP, Study Director — Shaheed Zulfiqar Ali Bhutto Medical University /PIMS
Locations (1):
- Shaheed Zulfiaqar Ali Bhutto Medical University, Islamabad, Federal Capital, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gautret P, Lagier JC, Parola P, Hoang VT, Meddeb L, Sevestre J, Mailhe M, Doudier B, Aubry C, Amrane S, Seng P, Hocquart M, Eldin C, Finance J, Vieira VE, Tissot-Dupont HT, Honore S, Stein A, Million M, Colson P, La Scola B, Veit V, Jacquier A, Deharo JC, Drancourt M, Fournier PE, Rolain JM, Brouqui P, Raoult D. Clinical and microbiological effect of a combination of hydroxychloroquine and azithromycin in 80 COVID-19 patients with at least a six-day follow up: A pilot observational study. Travel Med Infect Dis. 2020 Mar-Apr;34:101663. doi: 10.1016/j.tmaid.2020.101663. Epub 2020 Apr 11. PMID 32289548
- [Background] Mack HG. Hydroxychloroquine use during the COVID-19 pandemic 2020. Aust J Gen Pract. 2020 Apr 14;49. doi: 10.31128/AJGP-COVID-08. PMID 32294807
- [Background] Xiang YT, Jin Y, Wang Y, Zhang Q, Zhang L, Cheung T. Tribute to health workers in China: A group of respectable population during the outbreak of the COVID-19. Int J Biol Sci. 2020 Mar 15;16(10):1739-1740. doi: 10.7150/ijbs.45135. eCollection 2020. PMID 32226292
- [Background] Khan S, Siddique R, Ali A, Bai Q, Li Z, Li H, Shereen MA, Xue M, Nabi G. The spread of novel coronavirus has created an alarming situation worldwide. J Infect Public Health. 2020 Apr;13(4):469-471. doi: 10.1016/j.jiph.2020.03.005. Epub 2020 Apr 2. No abstract available. PMID 32247752